CLINICAL TRIAL: NCT00005147
Title: Epidemiology of Atherosclerosis
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1018; R01HL024489 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2000-04

CONDITIONS: Atherosclerosis; Cardiovascular Diseases; Heart Diseases; Coronary Arteriosclerosis
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases; Heart Diseases; Coronary Artery Disease

SUMMARY:
To determine the role of genetic factors in predicting resistance and susceptibility to coronary artery disease.

DETAILED DESCRIPTION:
BACKGROUND:

Coronary artery disease appears to be a consequence of the interaction between an individual's genotype and exposure to environmental factors. Genetic information has the potential to contribute to the identification of families and individuals with a biological predisposition for developing coronary artery disease. Although numerous studies have suggested the possibility of a link between polymorphic genetic variation and coronary heart disease, it has not been possible to use any single genetic locus or combination of loci to establish a person's risk except for the case of familial hypercholesterolemia.

Apolipoproteins play a critical role in regulating cellular uptake of lipoproteins by specific receptors, regulating the activities of lipoprotein lipase and lecithin-cholesterol acyl transferase, and in the indirect regulation of the intracellular enzymes, acyl-cholesterol acyl transferase and HMG Co-A reductase. This study provided insight into the role of environmental and genetic effects on phenotypic variation of the individual components of the molecules of lipid metabolism as well as on the relationships between components.

Previous studies conducted under this grant include: the relationship between quantitative levels of apo A-I and coronary artery disease as defined by coronary angiography; the effects of exercise, alcohol, obesity, and pregnancy on apo A-I levels; the relationship between apo A-I and HDL levels in children and the mode of inheritance of apo A-I levels in pedigrees in the Rochester, Minnesota community; and characterization of the antigenic structure of apolipoproteins in coronary artery disease.

DESIGN NARRATIVE:

Subjects for the study were drawn from the Rochester Family Heart Study which initiated recruitment for the family study in January 1985. In 31 months of recruitment, 443 households were contacted and 300 agreed to participate. In August 1987 all individuals identified by these households had completed their clinic visits providing 1,999 physical exams. The 300 households yielded 276 three and four generation pedigrees with 593 parents, 598 grandparents, 14 great-grandparents, and 854 children. Disease information was obtained from medical records for an additional 400 grandparents. In 1988 an additional 2,100 individual members of 300 families were surveyed.

Medical records and death certificates were reviewed to evaluate coronary artery disease endpoints in all adults members of the pedigrees. Clinical data collected included: a history of symptoms of coronary artery disease, arteriosclerosis obliterans, cerebrovascular disease or surgery for these diseases; smoking; medication; history of genetic relationships. Measurements were made of cholesterol, triglycerides, HDL and LDL cholesterol, apo A-I, apo A-II, apo E, apo C-III, apo C-II, apo B, apo Lp(a), LDL apo B, HDL apo E, and DNA extraction. Lipid, lipoprotein, and apolipoprotein phenotypes and the restriction fragment length polymorphisms (RFLP) were measured in candidate genes for coronary artery disease. Genetic and phenotype analyses were conducted at the University of Michigan. The RFLP and apolipoprotein isotyping analyses were conducted at the University of Pittsburgh. RFLP analysis and LDL receptor and A-I gene analysis were conducted at Charing Cross Medical Center in London, England.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1979-09; Study Completion 1991-06 (Actual)

REFERENCES:
- [Background] Mailly F, Moll P, Kottke BA, Kamboh MI, Humphries SE, Ferrell RE. Estimation of the frequency of isoform-genotype discrepancies at the apolipoprotein E locus in heterozygotes for the isoforms. Genet Epidemiol. 1992;9(4):239-48. doi: 10.1002/gepi.1370090403. PMID 1398044
- [Background] Reilly SL, Ferrell RE, Kottke BA, Kamboh MI, Sing CF. The gender-specific apolipoprotein E genotype influence on the distribution of lipids and apolipoproteins in the population of Rochester, MN. I. Pleiotropic effects on means and variances. Am J Hum Genet. 1991 Dec;49(6):1155-66. PMID 1842218
- [Background] Kottke BA, Moll PP, Michels VV, Weidman WH. Levels of lipids, lipoproteins, and apolipoproteins in a defined population. Mayo Clin Proc. 1991 Dec;66(12):1198-208. doi: 10.1016/s0025-6196(12)62470-7. PMID 1749288
- [Background] Kamboh MI, Ferrell RE, Kottke BA. Expressed hypervariable polymorphism of apolipoprotein (a). Am J Hum Genet. 1991 Nov;49(5):1063-74. PMID 1928089
- [Background] Kaprio J, Ferrell RE, Kottke BA, Kamboh MI, Sing CF. Effects of polymorphisms in apolipoproteins E, A-IV, and H on quantitative traits related to risk for cardiovascular disease. Arterioscler Thromb. 1991 Sep-Oct;11(5):1330-48. doi: 10.1161/01.atv.11.5.1330. PMID 1911720
- [Background] Turner ST, Michels VV. Sodium-lithium countertransport and hypertension in Rochester, Minnesota. Hypertension. 1991 Aug;18(2):183-90. doi: 10.1161/01.hyp.18.2.183. PMID 1885226
- [Background] Perusse L, Moll PP, Sing CF. Evidence that a single gene with gender- and age-dependent effects influences systolic blood pressure determination in a population-based sample. Am J Hum Genet. 1991 Jul;49(1):94-105. PMID 2063879
- [Background] Crews DE, Kamboh MI, Bindon JR, Ferrell RE. Genetic studies of human apolipoproteins. XVII: Population genetics of apolipoprotein polymorphisms in American Samoa. Am J Phys Anthropol. 1991 Feb;84(2):165-70. doi: 10.1002/ajpa.1330840206. PMID 2021192
- [Background] Kamboh MI, Weiss KM, Ferrell RE. Genetic studies of human apolipoproteins. XVI. APOE polymorphism and cholesterol levels in the Mayans of the Yucatan Peninsula, Mexico. Clin Genet. 1991 Jan;39(1):26-32. doi: 10.1111/j.1399-0004.1991.tb02981.x. PMID 1997212
- [Background] Kamboh MI, Ferrell RE. Genetic studies of human apolipoproteins. XV. An overview of IEF immunoblotting methods to screen apolipoprotein polymorphisms. Hum Hered. 1990;40(4):193-207. doi: 10.1159/000153931. PMID 2199367
- [Background] Ferrell RE, Kamboh MI, Majumder PP, Valdez R, Weiss KM. Genetic studies of human apolipoproteins. XIII. Quantitative polymorphism of apolipoprotein C-III in the Mayans of the Yucatan Peninsula. Hum Hered. 1990;40(3):127-35. doi: 10.1159/000153919. PMID 2365371
- [Background] Eichner JE, Kuller LH, Ferrell RE, Meilahn EN, Kamboh MI. Phenotypic effects of apolipoprotein structural variation on lipid profiles. III. Contribution of apolipoprotein E phenotype to prediction of total cholesterol, apolipoprotein B, and low density lipoprotein cholesterol in the healthy women study. Arteriosclerosis. 1990 May-Jun;10(3):379-85. doi: 10.1161/01.atv.10.3.379. PMID 2344296
- [Background] Kamboh MI, Kelly LJ, Ferrell RE. Genetic studies of human apolipoproteins: XIV. A simple agarose isoelectric focusing gel method for apolipoprotein E phenotyping. Electrophoresis. 1990 Apr;11(4):314-8. doi: 10.1002/elps.1150110408. PMID 2340826
- [Background] Rebbeck TR, Turner ST, Sing CF. Sodium-lithium countertransport genotype and the probability of hypertension in adults. Hypertension. 1993 Oct;22(4):560-8. doi: 10.1161/01.hyp.22.4.560. PMID 8406661
- [Background] Bren ND, Rastogi A, Kottke BA. Quantification of human plasma apolipoproteins C-I, C-II, and C-III by radioimmunoassays. Mayo Clin Proc. 1993 Jul;68(7):657-64. doi: 10.1016/s0025-6196(12)60601-6. PMID 8350639
- [Background] Pettitt DJ, Moll PP, Knowler WC, Mott DM, Nelson RG, Saad MF, Bennett PH, Kottke BA. Insulinemia in children at low and high risk of NIDDM. Diabetes Care. 1993 Apr;16(4):608-15. doi: 10.2337/diacare.16.4.608. PMID 8462388
- [Background] Maciejko JJ, Holmes DR, Kottke BA, Zinsmeister AR, Dinh DM, Mao SJ. Apolipoprotein A-I as a marker of angiographically assessed coronary-artery disease. N Engl J Med. 1983 Aug 18;309(7):385-9. doi: 10.1056/NEJM198308183090701. PMID 6410239
- [Background] Moll PP, Sing CF, Weidman WH, Gordon H, Ellefson RD, Hodgson PA, Kottke BA. Total cholesterol and lipoproteins in school children: prediction of coronary heart disease in adult relatives. Circulation. 1983 Jan;67(1):127-34. doi: 10.1161/01.cir.67.1.127. PMID 6847791
- [Background] Moll PP, Berry TD, Weidman WH, Ellefson R, Gordon H, Kottke BA. Detection of genetic heterogeneity among pedigrees through complex segregation analysis: an application to hypercholesterolemia. Am J Hum Genet. 1984 Jan;36(1):197-211. PMID 6607671
- [Background] Moll PP, Sing CF, Lussier-Cacan S, Davignon J. An application of a model for a genotype-dependent relationship between a concomitant (age) and a quantitative trait (LDL cholesterol) in pedigree data. Genet Epidemiol. 1984;1(4):301-14. doi: 10.1002/gepi.1370010403. PMID 6544242
- [Background] Kottke BA: The Role of Apolipoproteins A-I and A-II in Atherogenesis and Coronary Heart Disease: Clinical Measurements of Apolipoproteins. Perspect Lipid Disorders, 2:4-11, 1984
- [Background] Sing CF, Boerwinkle E, Moll PP. Strategies for elucidating the phenotypic and genetic heterogeneity of a chronic disease with a complex etiology. Prog Clin Biol Res. 1985;194:39-66. PMID 3906666
- [Background] Sing CF, Davignon J. Role of the apolipoprotein E polymorphism in determining normal plasma lipid and lipoprotein variation. Am J Hum Genet. 1985 Mar;37(2):268-85. PMID 3985008
- [Background] Sing CF et al: Apolipoproteins and Cardiovascular Risk: Genetics and Epidemiology. Ann Biol Clin, 43:411-417, 1985
- [Background] Sing CF, Boerwinkle E, Turner ST. Genetics of primary hypertension. Clin Exp Hypertens A. 1986;8(4-5):623-51. doi: 10.3109/10641968609046580. PMID 3530548
- [Background] Kottke BA: Perspectives in Medicine; Apolipoprotein Markers for Coronary Artery Diseases - A Dissenting View. Drug Ther, 16:151-171, 1986
- [Background] Boerwinkle E, Sing CF. Bias of the contribution of single-locus effects to the variance of a quantitative trait. Am J Hum Genet. 1986 Jul;39(1):137-44. PMID 3463204
- [Background] Moll PP, Sing CF, Williams RR, Mao SJ, Kottke BA. The genetic determination of plasma apolipoprotein A-I levels measured by radioimmunoassay: a study of high-risk pedigrees. Am J Hum Genet. 1986 Mar;38(3):361-72. PMID 3082191
- [Background] Boehnke M, Moll PP, Lange K, Weidman WH, Kottke BA. Univariate and bivariate analyses of cholesterol and triglyceride levels in pedigrees. Am J Med Genet. 1986 Mar;23(3):775-92. doi: 10.1002/ajmg.1320230306. PMID 3953676
- [Background] Boerwinkle E, Chakraborty R, Sing CF. The use of measured genotype information in the analysis of quantitative phenotypes in man. I. Models and analytical methods. Ann Hum Genet. 1986 May;50(2):181-94. doi: 10.1111/j.1469-1809.1986.tb01037.x. PMID 3435047
- [Background] Kottke BA, Zinsmeister AR, Holmes DR Jr, Kneller RW, Hallaway BJ, Mao SJ. Apolipoproteins and coronary artery disease. Mayo Clin Proc. 1986 May;61(5):313-20. doi: 10.1016/s0025-6196(12)61947-8. PMID 3702492
- [Background] Hurt RD, Briones ER, Offord KP, Patton JG, Mao SJ, Morse RM, Kottke BA. Plasma lipids and apolipoprotein A-I and A-II levels in alcoholic patients. Am J Clin Nutr. 1986 Apr;43(4):521-9. doi: 10.1093/ajcn/43.4.521. PMID 3962905
- [Background] Badimon JJ, Kottke BA, Chen TC, Chan L, Mao SJ. Quantification and immunolocalization of apolipoprotein E in experimental atherosclerosis. Atherosclerosis. 1986 Jul;61(1):57-66. doi: 10.1016/0021-9150(86)90113-9. PMID 3730054
- [Background] Au YP, Hallaway BJ, Kottke BA. Use of a quality-control plasma sample to decrease interassay variation in radioimmunoassays of apolipoprotein A-I. Clin Chem. 1986 Jul;32(7):1394-7. PMID 3087660
- [Background] Au YP, Bren ND, Kottke BA. A rapid apolipoprotein E radioimmunoassay using solid-phase staphylococcus protein. Use of pooled plasma as a secondary standard. Biochem Biophys Res Commun. 1986 Jul 16;138(1):455-62. doi: 10.1016/0006-291x(86)90302-5. PMID 3091017
- [Background] Kottke BA: Hyperlipoproteinemia. The Case for Individualized Care. Consultant, 26:160-169, 1986
- [Background] Boerwinkle E, Visvikis S, Welsh D, Steinmetz J, Hanash SM, Sing CF. The use of measured genotype information in the analysis of quantitative phenotypes in man. II. The role of the apolipoprotein E polymorphism in determining levels, variability, and covariability of cholesterol, betalipoprotein, and triglycerides in a sample of unrelated individuals. Am J Med Genet. 1987 Jul;27(3):567-82. doi: 10.1002/ajmg.1320270310. PMID 3631131
- [Background] Templeton AR, Boerwinkle E, Sing CF. A cladistic analysis of phenotypic associations with haplotypes inferred from restriction endonuclease mapping. I. Basic theory and an analysis of alcohol dehydrogenase activity in Drosophila. Genetics. 1987 Oct;117(2):343-51. doi: 10.1093/genetics/117.2.343. PMID 2822535
- [Background] Boerwinkle E, Sing CF. The use of measured genotype information in the analysis of quantitative phenotypes in man. III. Simultaneous estimation of the frequencies and effects of the apolipoprotein E polymorphism and residual polygenetic effects on cholesterol, betalipoprotein and triglyceride levels. Ann Hum Genet. 1987 Jul;51(3):211-26. doi: 10.1111/j.1469-1809.1987.tb00874.x. PMID 3688836
- [Background] Sing CF, Boerwinkle EA. Genetic architecture of inter-individual variability in apolipoprotein, lipoprotein and lipid phenotypes. Ciba Found Symp. 1987;130:99-127. doi: 10.1002/9780470513507.ch7. PMID 3327665
- [Background] Boehnke M, Moll PP, Kottke BA, Weidman WH. Partitioning the variability of fasting plasma glucose levels in pedigrees. Genetic and environmental factors. Am J Epidemiol. 1987 Apr;125(4):679-89. doi: 10.1093/oxfordjournals.aje.a114581. PMID 3826046
- [Background] Sing CF et al: Characterization of Genes Affecting Quantitative Traits in Humans. Proceedings Second International Conference on Quantitative Genetics, B. Weir (Ed.) Sinauer. In press, 1987
- [Background] Davignon J, Gregg RE, Sing CF. Apolipoprotein E polymorphism and atherosclerosis. Arteriosclerosis. 1988 Jan-Feb;8(1):1-21. doi: 10.1161/01.atv.8.1.1. PMID 3277611
- [Background] Lavie CJ, Gau GT, Squires RW, Kottke BA. Management of lipids in primary and secondary prevention of cardiovascular diseases. Mayo Clin Proc. 1988 Jun;63(6):605-21. doi: 10.1016/s0025-6196(12)64891-5. PMID 3287024
- [Background] Moll PP, Michels VV, Weidman WH, Kottke BA. Genetic determination of plasma apolipoprotein AI in a population-based sample. Am J Hum Genet. 1989 Jan;44(1):124-39. PMID 2491774
- [Background] Kaprio J, Ferrell RE, Kottke BA, Sing CF. Smoking and reverse cholesterol transport: evidence for gene-environment interaction. Clin Genet. 1989 Oct;36(4):266-8. doi: 10.1111/j.1399-0004.1989.tb03201.x. No abstract available. PMID 2509115
- [Background] Boehnke M, Moll PP. Identifying pedigrees segregating at a major locus for a quantitative trait: an efficient strategy for linkage analysis. Am J Hum Genet. 1989 Feb;44(2):216-24. PMID 2912068
- [Background] Turner ST, Weidman WH, Michels VV, Reed TJ, Ormson CL, Fuller T, Sing CF. Distribution of sodium-lithium countertransport and blood pressure in Caucasians five to eighty-nine years of age. Hypertension. 1989 Apr;13(4):378-91. doi: 10.1161/01.hyp.13.4.378. PMID 2925236
- [Background] Hasstedt SJ, Moll PP. Estimation of genetic model parameters: variables correlated with a quantitative phenotype exhibiting major locus inheritance. Genet Epidemiol. 1989;6(2):319-32. doi: 10.1002/gepi.1370060203. PMID 2721927
- [Background] Carlson TL, Kottke BA. Effect of 25-hydroxycholesterol and bile acids on the regulation of cholesterol metabolism in Hep G2 cells. Biochem J. 1989 Nov 15;264(1):241-7. doi: 10.1042/bj2640241. PMID 2513806
- [Background] Kottke BA, Friedlaender JS, Zerba KE, Sing CF. Lipid and apolipoprotein levels in six Solomon Island societies differ from those in a U.S. white population. Am J Phys Anthropol. 1990 Apr;81(4):483-91. doi: 10.1002/ajpa.1330810405. PMID 2110417
- [Background] Reilly SL, Kottke BA, Sing CF. The effects of generation and gender on the joint distributions of lipid and apolipoprotein phenotypes in the population at large. J Clin Epidemiol. 1990;43(9):921-40. doi: 10.1016/0895-4356(90)90076-2. PMID 2213081
- [Background] Sing CF, Haviland MB, Zerba KE, Templeton AR. Application of cladistics to the analysis of genotype-phenotype relationships. Eur J Epidemiol. 1992 May;8 Suppl 1:3-9. doi: 10.1007/BF00145343. PMID 1354623
- [Background] Reilly SL, Ferrell RE, Kottke BA, Sing CF. The gender-specific apolipoprotein E genotype influence on the distribution of plasma lipids and apolipoproteins in the population of Rochester, Minnesota. II. Regression relationships with concomitants. Am J Hum Genet. 1992 Dec;51(6):1311-24. PMID 1463013
- [Background] Hallaway BJ, Rastogi A, Kottke BA. Apolipoprotein B quantified by particle-concentration fluorescence immunoassay. Clin Chem. 1992 Dec;38(12):2387-91. PMID 1458572
- [Background] Turner ST, Rebbeck TR, Sing CF. Sodium-lithium countertransport and probability of hypertension in Caucasians 47 to 89 years old. Hypertension. 1992 Dec;20(6):841-50. doi: 10.1161/01.hyp.20.6.841. PMID 1452301
- [Background] Sing CF, Moll PP. Genetics of atherosclerosis. Annu Rev Genet. 1990;24:171-87. doi: 10.1146/annurev.ge.24.120190.001131. No abstract available. PMID 2088166